CLINICAL TRIAL: NCT03421730
Title: A Single-dose, Open-label, Randomized, Incomplete Block Design Trial to Characterize the Pharmacokinetics of VR647 Inhalation Suspension Delivered by the VR647 Inhalation System and Single Doses of Budesonide Delivered by a Conventional Jet Nebulizer in Pediatric Subjects Aged 4 to 8 Years With Wheezing, Reactive Airway Disease or Mild Asthma
Brief Title: A Study of the Pharmacokinetics, Safety and Tolerability of Single Doses of VR647 Inhalation Suspension Administered Using the VR647 Inhalation System in Children With Wheezing, Reactive Airway Disease or Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vectura Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VR647/1/002
Record Dates: First submitted 2018-01-12; First posted 2018-02-05 (Actual); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Wheezing; Reactive Airway Disease; Mild Asthma
Keywords: mild asthma; budesonide; nebulizer; pediatric; pharmacokinetics
MeSH Terms: conditions — Respiratory Sounds; Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Intervention Model Description: This is an open label, randomized, balanced, incomplete block design trial. Eligible subjects will be randomized to 1 of 12 treatment sequences (A,B), (A,C), (A,D), (B,A), (B,C), (B,D), (C,A), (C,B), (C,D), (D,A), (D,B) or (D,C), corresponding to the following treatment regimens:
  * (A) 5 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System
  * (B) 10 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System
  * (C) 20 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System
  * (D) 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer nebulized to empty
  The treatment period comprises 2 dosing visits. Each subject will receive their first treatment regimen during Visit 2 and their second treatment regimen during Visit 3.
Masking Description: This is an open label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- AB - VR647 5 breaths, then VR647 10 breaths (Experimental): 5 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 10 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System
- AC - VR647 5 breaths, then VR647 20 breaths (Experimental): 5 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 20 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System
- AD - VR647 5 breaths, then Pulmicort (Experimental): 5 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 1 mg/2 mL Pulmicort Respules delivered by the conventional jet nebulizer nebulized to empty
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer
- BA - VR647 10 breaths, then VR647 5 breaths (Experimental): 10 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 5 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System
- BC - VR647 10 breaths, then VR647 20 breaths (Experimental): 10 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 20 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System
- BD - VR647 10 breaths, then Pulmicort (Experimental): 10 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 1 mg/2 mL Pulmicort Respules delivered by the conventional jet nebulizer nebulized to empty
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer
- CA - VR647 20 breaths, then VR647 5 breaths (Experimental): 20 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 5 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System
- CB - VR647 20 breaths, then VR647 10 breaths (Experimental): 20 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 10 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System
- CD - VR647 20 breaths, then Pulmicort (Experimental): 20 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System followed by 1 mg/2 mL Pulmicort Respules delivered by the conventional jet nebulizer nebulized to empty
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer
- DA - Pulmicort, then VR647 5 breaths (Experimental): 1 mg/2 mL Pulmicort Respules delivered by the conventional jet nebulizer nebulized to empty followed by 5 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer
- DB - Pulmicort, then VR647 10 breaths (Experimental): 1 mg/2 mL Pulmicort Respules delivered by the conventional jet nebulizer nebulized to empty followed by 10 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer
- DC - Pulmicort, then VR647 20 breaths (Experimental): 1 mg/2 mL Pulmicort Respules delivered by the conventional jet nebulizer nebulized to empty followed by 20 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  Interventions: Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System; Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer

INTERVENTIONS:
Combination Product: VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System — The VR647 Inhalation System consists of the VR647 Inhalation System 1 control unit, a VR647 nebulizer handset, a mouthpiece and VR647 Smart Cards designed specifically for this trial.
Combination Product: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer — Commercial Pulmicort Respules (budesonide inhalation suspension 1 mg/2 mL) delivered by a conventional jet nebulizer operated to sputtering.
  Arms: AD - VR647 5 breaths, then Pulmicort; BD - VR647 10 breaths, then Pulmicort; CD - VR647 20 breaths, then Pulmicort; DA - Pulmicort, then VR647 5 breaths; DB - Pulmicort, then VR647 10 breaths; DC - Pulmicort, then VR647 20 breaths

SUMMARY:
The primary objective of this study is to evaluate budesonide levels in the blood following inhalation of single doses of VR647 Inhalation Suspension in children with wheezing, reactive airway disease or mild asthma using a nebulizer, the VR647 Inhalation System. Secondary objectives include the evaluation of the safety and tolerability of VR647 Inhalation Suspension administered using the VR647 Inhalation System.

The study consists of four visits; a screening visit (Visit 1), two dosing days (Visits 2 and 3) and a follow-up visit (Visit 4). On each dosing day a single dose of treatment will be administered. Treatment allocation at Visits 2 and 3 is determined by a balanced incomplete block design.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or pre-menarchal female subjects.
* Aged 4 to 8 years, inclusive.
* Diagnosis of wheezing, reactive airway disease or mild asthma confirmed by a physician at least 3 months prior to screening.
* Wheezing, reactive airway disease or mild asthma controlled by intermittent or regular non-steroidal medications commonly used for asthma, such as short-acting β2-agonists (SABAs) or leukotriene receptor antagonists (LTRAs), for a minimum of 28 days prior to the Screening Visit.
* Body weight ≥15 kg.
* Subject is able to demonstrate the ability to use the VR647 Inhalation System and the conventional jet nebulizer effectively during training.

Key Exclusion Criteria:

* Clinically relevant abnormality or medical condition (other than wheezing, reactive airway disease or mild asthma) identified at the screening assessment that, in the opinion of the investigator, could interfere with the objectives of the trial or the safety of the subject. The sponsor's medical officer should be consulted in case of any doubt.
* Life-threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episodes.
* Subjects currently using long-acting β2-agonists.
* Use of the following prescription medications within 28 days prior to the first treatment day: corticosteroids by any route and drugs that inhibit cytochrome P450 3A4.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Burgess, MD, Study Director — Vectura Ltd
Locations (3):
- United States (3):
  - Vectura Study Site 0003, Colorado Springs, Colorado
  - Vectura Study Site 0002, Raleigh, North Carolina
  - Vectura Study Site 0001, Tulsa, Oklahoma

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventeen subjects were enrolled and randomized to 1 of 12 crossover treatment sequences AB, AC, AD, BA, BC, BD, CA, CB, CD, DA, DB or DC. However, data were analyzed (and presented) by individual treatment only (i.e. A, B, C and D), not per treatment sequence. Fifteen subjects received at least 1 study treatment; 13 subjects completed the trial.
Groups:
- AB - VR647 5 Breaths, Then VR647 10 Breaths: 5 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (A) followed by 10 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (B)
- AC - VR647 5 Breaths, Then VR647 20 Breaths: 5 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (A) followed by 20 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (C)
- AD - VR647 5 Breaths, Then Pulmicort: 5 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (A) followed by 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer nebulized to empty (D)
- BA - VR647 10 Breaths, Then VR647 5 Breaths: 10 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (B) followed by 5 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (A)
- BC - VR647 10 Breaths, Then VR647 20 Breaths: 10 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (B) followed by 20 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (C)
- BD - VR647 10 Breaths, Then Pulmicort: 10 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (B) followed by 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer nebulized to empty (D)
- CA - VR647 20 Breaths, Then VR647 5 Breaths: 20 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (C) followed by 5 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (A)
- CB - VR647 20 Breaths, Then VR647 10 Breaths: 20 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (C) followed by 10 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (B)
- CD - VR647 20 Breaths, Then Pulmicort: 20 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (C) followed by 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer nebulized to empty (D)
- DA - Pulmicort, Then VR647 5 Breaths: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer nebulized to empty (D) followed by 5 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (A)
- DB - Pulmicort, Then VR647 10 Breaths: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer nebulized to empty (D) followed by 10 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (B)
- DC - Pulmicort, Then VR647 20 Breaths: 1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer nebulized to empty (D) followed by 20 breaths of VR647 Inhalation Suspension delivered by the VR647 Inhalation System (C)
Period: First Intervention (Day 1, Visit 2)
Arm/Group | AB - VR647 5 Breaths, Then VR647 10 Breaths | AC - VR647 5 Breaths, Then VR647 20 Breaths | AD - VR647 5 Breaths, Then Pulmicort | BA - VR647 10 Breaths, Then VR647 5 Breaths | BC - VR647 10 Breaths, Then VR647 20 Breaths | BD - VR647 10 Breaths, Then Pulmicort | CA - VR647 20 Breaths, Then VR647 5 Breaths | CB - VR647 20 Breaths, Then VR647 10 Breaths | CD - VR647 20 Breaths, Then Pulmicort | DA - Pulmicort, Then VR647 5 Breaths | DB - Pulmicort, Then VR647 10 Breaths | DC - Pulmicort, Then VR647 20 Breaths
Started | 1 | 3 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 (Two subjects withdrew without receiving treatment with either A or C.) | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by subject or legal guardian | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (Days 4 to 10)
Arm/Group | AB - VR647 5 Breaths, Then VR647 10 Breaths | AC - VR647 5 Breaths, Then VR647 20 Breaths | AD - VR647 5 Breaths, Then Pulmicort | BA - VR647 10 Breaths, Then VR647 5 Breaths | BC - VR647 10 Breaths, Then VR647 20 Breaths | BD - VR647 10 Breaths, Then Pulmicort | CA - VR647 20 Breaths, Then VR647 5 Breaths | CB - VR647 20 Breaths, Then VR647 10 Breaths | CD - VR647 20 Breaths, Then Pulmicort | DA - Pulmicort, Then VR647 5 Breaths | DB - Pulmicort, Then VR647 10 Breaths | DC - Pulmicort, Then VR647 20 Breaths
Started | 1 | 1 | 1 | 1 | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 (Two subjects withdrew after receiving treatment with B but before receiving treatment with C.) | 1 | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by subject or legal guardian | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (Day 8±3, Visit 3)
Arm/Group | AB - VR647 5 Breaths, Then VR647 10 Breaths | AC - VR647 5 Breaths, Then VR647 20 Breaths | AD - VR647 5 Breaths, Then Pulmicort | BA - VR647 10 Breaths, Then VR647 5 Breaths | BC - VR647 10 Breaths, Then VR647 20 Breaths | BD - VR647 10 Breaths, Then Pulmicort | CA - VR647 20 Breaths, Then VR647 5 Breaths | CB - VR647 20 Breaths, Then VR647 10 Breaths | CD - VR647 20 Breaths, Then Pulmicort | DA - Pulmicort, Then VR647 5 Breaths | DB - Pulmicort, Then VR647 10 Breaths | DC - Pulmicort, Then VR647 20 Breaths
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 17 subjects were enrolled. However, 2 subjects withdrew from the study prior to treatment with the first intervention. As baseline characteristics were not reported for these two subjects, the overall number of baseline participants was 15 subjects.
Groups:
- Overall Treatment: Baseline measures were not analysed by arm or comparison group, so they are presented for the total number of subjects enrolled in the study who received at least one dose of treatment.
Arm/Group | Overall Treatment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: months] | 82.6 (14.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: AUClast of Plasma Budesonide (VR647 Inhalation Suspension Delivered by the VR647 Inhalation System or Pulmicort Respules Delivered by a Conventional Jet Nebulizer).
Description: AUClast is the area under the plasma concentration-time curve, from time 0 to the time of the last measurable concentration (Clast).
Time Frame: Pre-dose, and at 20 minutes, 40 minutes, 1.5, 3, 4, 6 and 8 hours after start of nebulization on Day 1 (Visit 2) and Day 8 (Visit 3).
Population: Pharmacokinetic set included 13 (76%) subjects.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Groups:
- A - 5 Breaths VR647: 5 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System: The VR647 Inhalation System consists of the VR647 Inhalation System 1 control unit, a VR647 nebulizer handset, a mouthpiece and VR647 Smart Cards designed specifically for this trial.
- B - 10 Breaths VR647: 10 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System: The VR647 Inhalation System consists of the VR647 Inhalation System 1 control unit, a VR647 nebulizer handset, a mouthpiece and VR647 Smart Cards designed specifically for this trial.
- C - 20 Breaths VR647: 20 breaths of the VR647 Inhalation Suspension 1 mg/2 mL delivered by the VR647 Inhalation System
  VR647 Inhalation Suspension (budesonide) 1 mg/2 mL delivered by the VR647 Inhalation System: The VR647 Inhalation System consists of the VR647 Inhalation System 1 control unit, a VR647 nebulizer handset, a mouthpiece and VR647 Smart Cards designed specifically for this trial.
- D - Pulmicort: 1 mg/2 mL Pulmicort Respules delivered by the conventional jet nebulizer nebulized to empty
  1 mg/2 mL Pulmicort Respules delivered by a conventional jet nebulizer: Commercial Pulmicort Respules (budesonide inhalation suspension 1 mg/2 mL) delivered by a conventional jet nebulizer operated to sputtering.
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 6 | 7 | 6 | 5
pg*hr/mL | 120.7 (20.498) | 327.5 (119.49) | 759.5 (311.79) | 1357 (564.06)
Statistical Analysis 1: Comparison: A - 5 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 8.69 — A: n=6; D: n=5; The intra-subject coefficient of variation was 25.33%
Statistical Analysis 2: Comparison: B - 10 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 28.18 — B: n=6, D: n=5; The intra-subject coefficient of variation was 25.33%
Statistical Analysis 3: Comparison: C - 20 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 59.51 — C: n=6, D: n=5; The intra-subject coefficient of variation was 25.33%

2. Primary Outcome: AUCinf of Plasma Budesonide (VR647 Inhalation Suspension Delivered by the VR647 Inhalation System or Pulmicort Respules Delivered by a Conventional Jet Nebulizer).
Description: AUCinf is the area under the plasma concentration-time curve, from time 0 extrapolated to infinity. AUCinf is calculated as the sum of AUClast plus the ratio of the last measurable plasma concentration (Clast) to the elimination rate constant (λz).
Time Frame: as for outcome 1
Population: Pharmacokinetic set included 13 (76%) subjects.
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 4 | 6 | 5 | 4
pg*hr/mL | 138.3 (25.189) | 326.2 (116.09) | 737.1 (313.27) | 1492 (707.99)
Statistical Analysis 1: Comparison: A - 5 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 13.35 — A: n=4, D: n=4; The intra-subject coefficient of variation was 22.05%
Statistical Analysis 2: Comparison: B - 10 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 35.97 — B: n=4, D: n=4; The intra-subject coefficient of variation was 22.05%
Statistical Analysis 3: Comparison: C - 20 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 76.98 — C: n=4, D: n=4; The intra-subject coefficient of variation was 22.05%

3. Primary Outcome: Cmax of Plasma Budesonide (VR647 Inhalation Suspension Delivered by the VR647 Inhalation System or Pulmicort Respules Delivered by a Conventional Jet Nebulizer).
Description: Cmax is the maximum observed concentration.
Time Frame: as for outcome 1
Population: Pharmacokinetic set included 13 (76%) subjects.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 6 | 7 | 6 | 5
pg/mL | 71.25 (9.5776) | 179.7 (79.442) | 390.3 (178.07) | 601.8 (405.32)
Statistical Analysis 1: Comparison: A - 5 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 9.55 — A: n=6, D: n=5; The intra-subject coefficient of variation was 33.04%
Statistical Analysis 2: Comparison: B - 10 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 32.42 — B: n=6, D: n=5; The intra-subject coefficient of variation was 33.04%
Statistical Analysis 3: Comparison: C - 20 Breaths VR647 vs D - Pulmicort; Test type: Other; Geometric mean ratio (%) = 59.75 — C: n=6, D: n=5; The intra-subject coefficient of variation was 33.04%

4. Primary Outcome: Tmax of Plasma Budesonide (VR647 Inhalation Suspension Delivered by the VR647 Inhalation System or Pulmicort Respules Delivered by a Conventional Jet Nebulizer).
Description: Tmax is the time to reach Cmax.
Time Frame: as for outcome 1
Population: Pharmacokinetic set included 13 (76%) subjects.
Measure: Median (Full Range); unit: hours
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 6 | 7 | 6 | 5
hours | 0.3330 [0.317 to 0.367] | 0.3330 [0.317 to 0.350] | 0.3500 [0.300 to 0.700] | 0.3330 [0.333 to 0.367]

5. Primary Outcome: Tlast of Plasma Budesonide (VR647 Inhalation Suspension Delivered by the VR647 Inhalation System or Pulmicort Respules Delivered by a Conventional Jet Nebulizer).
Description: Tlast is the time of the last measurable concentration (Clast).
Time Frame: as for outcome 1
Population: Pharmacokinetic set included 13 (76%) subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 6 | 7 | 6 | 5
hours | 5.325 (1.6331) | 7.386 (0.9539) | 7.620 (0.7962) | 7.937 (0.0447)

6. Primary Outcome: T1/2 of Plasma Budesonide (VR647 Inhalation Suspension Delivered by the VR647 Inhalation System or Pulmicort Respules Delivered by a Conventional Jet Nebulizer).
Description: T1/2 is the apparent first-order terminal elimination half-life.
Time Frame: as for outcome 1
Population: Pharmacokinetic set included 13 (76%) subjects.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 4 | 6 | 5 | 4
hours | 1.703 (0.7005) | 1.991 (0.3587) | 2.059 (0.5895) | 2.200 (0.3300)

7. Secondary Outcome: Mean Modified Patient Satisfaction and Preference Questionnaire (PASAPQ) Total Score (Q1 to Q8).
Description: The PASAPQ is a validated multi-item measure of satisfaction and preference with inhaler devices. The modified PASAPQ consists of 10 questions. The first 8 questions generate the total score domain. Data from this questionnaire were listed by subject and summarized by treatment. The results from Questions 1 through 8 were added for each subject to generate the Total Score (n = Q1+Q2+Q3+Q4+Q5+Q6+Q7+Q8) and expressed as percentage of maximum total score (i.e., (n/56)*100). Questions 1 to 8 were answered using scores from 1 (i.e., very dissatisfied) to 7 (i.e., very satisfied).
Time Frame: Following dosing on Day 1 (Visit 2) and Day 8 (Visit 3).
Population: Safety set included 15 (88%) subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: percentage of maximum total score
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
percentage of maximum total score | 97.7 (3.95) | 95.8 (7.23) | 97.5 (3.56) | 88.6 (8.28)

8. Secondary Outcome: Mean Modified PASAPQ Performance Score
Description: The PASAPQ is a validated multi-item measure of satisfaction and preference with inhaler devices; it was originally a 15-item questionnaire, with performance assessed over 7 items. The modified PASAPQ (mPASAPQ) has 10 questions, including only 4 from the performance domain; the 3 questions not included were dropped from the mPASAPQ as they were not applicable to patient population and device under study. Questions 1, 2, 6, and 7 were assessed, covering satisfaction with nebulizer reliability, ease of inhalation, use and treatment time. Although specified in the protocol, the mPASAPQ performance score was not summarized in the efficacy analysis. The results for each question are presented below, however it was not considered appropriate to analyze the performance domain, as it is not possible to verify the validity of the questionnaire utilising only 4 of the original 7 questions. Questions were answered using scores from 1 (i.e., very dissatisfied) to 7 (i.e., very satisfied).
Time Frame: Following dosing on Day 1 (Visit 2) and Day 8 (Visit 3).
Population: Although specified in the protocol, mPASAPQ performance score wasn't summarized in the efficacy analysis as 3 questions were dropped from the PASAPQ that were not applicable. This change from the protocol-planned analysis was described in the SAP, finalized before DB lock. Individual scores for the 4 remaining performance questions are presented.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
scores on a scale
  Question 1 | 6.9 (0.38) | 6.6 (0.52) | 6.3 (0.82) | 6.4 (0.53)
  Question 2 | 6.9 (0.38) | 6.5 (0.76) | 7.0 (0.00) | 6.0 (1.15)
  Question 6 | 6.7 (0.49) | 6.6 (0.52) | 6.8 (0.41) | 6.1 (1.07)
  Question 7 | 7.0 (0.00) | 6.8 (0.71) | 7.0 (0.00) | 5.3 (1.60)

9. Secondary Outcome: Mean Modified PASAPQ Satisfaction Score (Q9).
Description: The PASAPQ is a validated multi-item measure of satisfaction and preference with inhaler devices. The modified PASAPQ consists of 10 questions. Question 9 asks for overall satisfaction with the device(s) used in the trial. Question 9 was answered using scores from 1 (i.e., very dissatisfied) to 7 (i.e., very satisfied).
Time Frame: Following dosing on Day 1 (Visit 2) and Day 8 (Visit 3).
Population: Safety set included 15 (88%) subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
scores on a scale | 6.9 (0.38) | 6.6 (0.74) | 6.8 (0.41) | 5.7 (0.95)

10. Secondary Outcome: Mean Modified PASAPQ Score Indicating Willingness to Continue With the Device (Q10).
Description: The PASAPQ is a validated multi-item measure of satisfaction and preference with inhaler devices. The modified PASAPQ consists of 10 questions. Question 10 asks about willingness to continue with the device(s) used in the trial. Parents/legal guardians were asked to indicate how willing they would be for their child to use the nebulizer used during the study, providing a number between 0 (unwilling) and 100 (willing).
Time Frame: Following dosing on Day 1 (Visit 2) and Day 8 (Visit 3).
Population: Safety set included 15 (88%) subjects who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
scores on a scale | 98.6 (3.78) | 93.5 (11.75) | 98.3 (4.08) | 77.3 (22.10)

11. Secondary Outcome: Changes in Vital Signs (Blood Pressure)
Description: Mean values for blood pressure from pre-dose to 0.5 hours post-dose.
Time Frame: Baseline to Day 1 0.5 hours post-dose
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
mm Hg
  Change in systolic blood pressure | -8.4 (8.40) | 9.0 (5.35) | 0.8 (4.67) | 4.4 (5.19)
  Change in diastolic blood pressure | -7.4 (13.60) | 2.1 (7.30) | -6.3 (12.93) | 1.9 (9.51)

12. Secondary Outcome: Changes in Vital Signs (Heart Rate)
Description: Mean values for heart rate from pre-dose to 0.5 hours post-dose.
Time Frame: Baseline to Day 1 0.5 hours post-dose
Measure: Mean (Standard Deviation); unit: change in beats per minute
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
change in beats per minute | 6.6 (9.86) | 2.6 (13.18) | 4.0 (11.30) | -2.6 (17.09)

13. Secondary Outcome: Changes in Vital Signs (Respiration Rate)
Description: Mean values for respiratory rate from pre-dose to 0.5 hours post-dose.
Time Frame: Baseline to Day 1 0.5 hours post-dose
Measure: Mean (Standard Deviation); unit: Change in breaths per minute
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
Change in breaths per minute | 0.0 (1.15) | 0.3 (0.71) | 0.3 (1.51) | 0.3 (0.76)

14. Secondary Outcome: Changes in Vital Signs (Temperature)
Description: Mean values for temperature from pre-dose to 0.5 hours post-dose.
Time Frame: Baseline to Day 1 0.5 hours post-dose
Measure: Mean (Standard Deviation); unit: Change in degrees Celsius
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
Change in degrees Celsius | 0.27 (0.373) | 0.04 (0.320) | 0.05 (0.207) | 0.14 (0.351)

15. Secondary Outcome: Changes in Physical Examination
Description: Physical examination data were listed. The number of participants with a change in physical examination status (i.e. from normal to abnormal, or from abnormal to normal) is presented below.
Time Frame: Visit 1, and Day 8 of Visit 3.
Measure: Count of Participants; unit: Participants
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Use of Concomitant Medications
Description: Number of subjects using concomitant medications.
Time Frame: Visit 1
Measure: Count of Participants; unit: Participants
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort
Number analyzed (Participants) | 7 | 8 | 6 | 7
Participants | 7 | 8 | 6 | 7

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and adverse device effects were monitored throughout the trial, until resolution. The total duration of participation for each subject was approximately 47 days, which included a 30-day screening period, two dosing visits with a washout period of 4 to 10 days between each dose, and a follow-up assessment approximately 7 days after last nebulization.
Description: Any changes from baseline (pre-dose value on Day 1) in vital signs and physical examination findings that were judged to be clinically significant were recorded as AEs.
Groups:
- Overall Treatment: The total number of subjects enrolled in the study who received at least one dose of treatment.
Arm/Group | A - 5 Breaths VR647 | B - 10 Breaths VR647 | C - 20 Breaths VR647 | D - Pulmicort | Overall Treatment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/6 | 0/7 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 0/6 | 0/7 | 0/15
Other Adverse Events (participants affected / at risk) | 1/7 | 1/8 | 1/6 | 0/7 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - 5 Breaths VR647 (N=7) | B - 10 Breaths VR647 (N=8) | C - 20 Breaths VR647 (N=6) | D - Pulmicort (N=7) | Overall Treatment (N=15)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication can be delayed for 60 days for Sponsor review and revisions/deletions can be required. Furthermore, a 6-month delay to publication can be required by the Sponsor in order to take steps to protect its proprietary information and/or intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT03421730/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT03421730/SAP_001.pdf